CLINICAL TRIAL: NCT00749216
Title: Multiple-Dose Safety in Japanese Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Solanezumab Safety Study in Japanese Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12025; H8A-JE-LZAK (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — solanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- QW (Experimental): IV infusion of 400mg once each week for 2 months
  Interventions: Drug: Solanezumab
- Q4W (Experimental): IV infusion of 400mg once every four weeks for 2 months
  Interventions: Drug: Solanezumab
- Q8W (Experimental): IV infusion of 400mg once every eight weeks for 2 months
  Interventions: Drug: Solanezumab

INTERVENTIONS:
Drug: Solanezumab
  Other Names: LY2062430

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of multiple dosing Solanezumab in subjects with mild-to-moderate AD in Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-fertile women, at least 50 years of age.(Women who are not surgically sterilized must be post-menopausal for at least 1 year.)
* Patients with mild to moderate AD by following disease diagnostic criteria

  * National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria
  * Modified Hachinski Ischemia Scale score of ≦ 4
  * Folstein Mini-Mental State Examination (MMSE) score of 15 through 26
  * Geriatric Depression Scale (GDS) score of ≦ 10 on the staff-administered short form

Exclusion Criteria:

* Patients who don't have a reliable caregiver who is in frequent contact with the patient, who will accompany the patient to the office and/or be available by telephone at designated times, and will monitor administration of prescribed medications.
* Patients who have an MRI or CT scan since the onset of symptoms of AD that is inconsistent with a diagnosis of AD.
* Patients who have received acetylcholinesterase inhibitors (AChEIs) or memantine for less than 4 months, or have less than 2 months of stable therapy on these treatments.
* Patients who have current serious or unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator or subinvestigator(s)'s opinion, could interfere with the analyses of safety and efficacy in this study.
* Patients who have a history within the last 5 years of a serious infectious disease affecting the brain (including neurosyphilis, meningitis, or encephalitis) or head trauma resulting in protracted loss of consciousness within the last 5 years, or multiple episodes of head trauma.
* Patients who have a history within the last 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal PSA post-resection.
* Patients who have allergies to humanized monoclonal antibodies.
* Patients who have a history within the last 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal PSA post-resection.
* Patients who have ECG abnormalities obtained that, in the opinion of the investigator, are clinically significant with regard to the subject's participation in the study, including QTc prolongation (Bazett's corrected QTc interval, QTcB; males >435 msec or females >455 msec) or abnormally wide QRS complexes (resulting from bundle-branch blocks, interventricular conduction delays, or pacemakers).
* Patients who have a current, required use or expected use of excluded drugs through the duration(These drugs include typical neuroleptics (antipsychotics). In addition, typical neuroleptics may not be taken within 4 weeks.
* Patients who are currently taking chronic medications that affect central nervous system (CNS) function, and are not dose-stabilized for at least 4 weeks.
* Patients who have a ventriculoperitoneal shunt or gamma globulin (IgG) therapy within the last year.
* Patients who have previously completed or withdrawn from this study or previous participation in any other study investigating active immunization against Aβ.
* Patients who have any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or cardiac pacemaker.
* Patients who weigh less than 40 kg.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months

SECONDARY OUTCOMES:
Changes in the extended ADAS-Cog stand for Alzheimer's Disease Assessment Scale-Cognitive subscale | 6 months
pharmacodynamic of Aβ1-40 and Aβ1-42 | 6 months
Pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com